CLINICAL TRIAL: NCT06453629
Title: A Randomized Controlled Study to Evaluate Social Skill Treatment Options in Children With Autism Using VR Technology
Brief Title: RCT to Evaluate Social Skills in Children With Autism Using VR Technology (SoCaVR)
Acronym: SoCaVR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Floreo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FLO-CL-2023-001
Record Dates: First submitted 2024-05-31; First posted 2024-06-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder; Social Communication
Keywords: Virtual Reality
MeSH Terms: conditions — Autism Spectrum Disorder; Communication

STUDY DESIGN:
Intervention Model Description: Experimental: Floreo VR- 12 week with follow up Active Comparator: VR Control- 12 week with ability to crossover or follow up Other: VR Control Crossover- 12 week of Floreo VR
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and their adult caregiver will be blinded. The Outcomes Assessor (Clinician) with the adult caregiver will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Floreo VR (Experimental): Floreo VR is a 12 week program
  Interventions: Device: Floreo VR
- VR Control (Active Comparator): VR Control is a 12 week program that matches the Floreo VR interactions
  Interventions: Device: VR Control
- VR Control Crossover (Other): For participants who opt in, they will run the 12 week Floreo VR program
  Interventions: Device: Floreo VR; Device: VR Control Crossover

INTERVENTIONS:
Device: Floreo VR — 12 week VR program to help children with ASD to reduce the core symptoms of Autism
  Arms: Floreo VR; VR Control Crossover
Device: VR Control — 12 week program administered in VR
  Arms: VR Control
Device: VR Control Crossover — If opt in, this group will crossover at the end of 12 weeks to the Floreo VR program
  Other Names: Crossover group
  Arms: VR Control Crossover

SUMMARY:
The goal of this randomized clinical trial is to compare and learn about Virtual Reality (VR) in children with autism/Autistic children.

The main question it aims to answer is:

• Does the Floreo VR clinical product show clinical improvement in autism symptoms?

Participants will engage the VR product for twice a week for twelve weeks.

They will be randomized to either the Floreo Clinical Product or a VR Control group experience.

Researchers will compare the two groups to see if there is an effect on learning specific skills and behaviors.

DETAILED DESCRIPTION:
The purpose of this study is to find out if Floreo's VR clinical program can help with autism symptoms such as social communication skills in autistic children. Recent advances in VR technology offers a new way to improve these types of skills in children with autism in an immersive and controlled environment.

Questionnaires answered by adult caregivers will be used to assess the child's behaviors during the time of treatment.

Clinician observations will also be conducted as a part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Five to eighteen years old (inclusive) at the time of consent
* Legal guardian is able and willing to properly sign and date informed consent indicating that they have been informed about the study and able to complete all visits [If age appropriate, an assent will also be administered to the participant to inform them of the study and give them an opportunity to proceed or decline]
* Verified diagnosis of ASD documented by a qualified clinician according to DSM-V criteria
* Receiving therapies at least two times per week in a clinic setting
* Participant is able to complete and pass the VR orientation screening

Exclusion Criteria:

* Significant medical condition(s) [examples listed below] or other circumstances which, in the opinion of the treating clinician, would preclude compliance with the protocol, adequate cooperation in the study, or may prevent the participant from safely participating in the study:
* Uncontrolled neurological conditions such as epilepsy, migraine
* Current disorders affecting balance, such as vertigo
* Primary sensory impairment such as blindness or deafness
* Eye movement impairment, such as strabismus
* Participants are enrolled in another clinical study
* Participants known to be pregnant
* Participation in this study is not in the best interest of the child, at the discretion of the treating clinician and the primary investigator.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Autism Impact Measure (AIM) | Baseline-12 weeks
  The primary objective of this study is to determine if administration of the Floreo VR compared to VR Control results in clinically significant improvement in autism symptoms as measured by the Autism Impact Measure (AIM) in the study participant population.

SECONDARY OUTCOMES:
Assessment of Functional Living Skills (AFLS) | Baseline-12 weeks
  Change from baseline to 12 weeks in scores on the subdomains of social skills and basic communications in the Assessment of Functional Living Skills (AFLS)
Child and Family Quality of Life (CFQL-2) | Baseline-12 weeks
  Change from baseline to 12 weeks in scores of the Child and Family Quality of Life (CFQL-2)
Assessment of Functional Living Skills (AFLS) | baseline, 16 weeks, 20 weeks, 24 weeks
  Change from 16, 20, 24 weeks in scores on the subdomains of social skills and basic communications in the Assessment of Functional Living Skills (AFLS)
Total Autism Impact Measure (AIM) Score | baseline, 16 weeks, 20 weeks, 24 weeks
  Responder rate at 16, 20, and 24 weeks for the Total AIM score
Child and Family Quality of Life (CFQL-2) | baseline, 16, 20, and 24 weeks
  Change from baseline to 24 weeks in scores on the subdomains of social skills and basic communications in the Assessment of Functional Living Skills (AFLS)

OTHER OUTCOMES:
Childhood Autism Rating Scale (CARS-2) | baseline, 12 weeks, 24 weeks
  Change from baseline,12, and 24 weeks in scores on the Childhood Autism Rating Scales-2 (CARS-2)
Floreo Skills Acquisition and Observations | baseline, 12 weeks, 24 weeks
  Floreo specific skills scores
Rate of Skills Acquisition | baseline, 12 weeks, 24 weeks
  Social Skills goals
Subdomain 1 of the Autism Impact Measure in Repetitive Behaviors | baseline, 12 weeks, 24 weeks
  Subdomain of the Autism Impact Measure in Repetitive Behaviors
Subdomain 2 of the Autism Impact Measure in Communications | baseline, 12 weeks, 24 weeks
  Subdomain of the Autism Impact Measure in Communications
Subdomain 3 of the Autism Impact Measure in Atypical Behavior | baseline, 12 weeks, 24 weeks
  Subdomain of the Autism Impact Measure in Atypical Behavior
Subdomain 4 of the Autism Impact Measure in Social Reciprocity | baseline, 12 weeks, 24 weeks
  Subdomain of the Autism Impact Measure in Social Reciprocity
Subdomain 5 of the Autism Impact Measure in Peer Interaction | baseline, 12 weeks, 24 weeks
  Subdomain of the Autism Impact Measure in Peer Interaction
Subdomain 6 of the Autism Impact Measure in questions not related to other subdomains | baseline, 12 weeks, 24 weeks
  Subdomain of the Autism Impact Measure in questions not related to other subdomains

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Goh, MD, Principal Investigator — Cortica
Locations (17):
- United States (17):
  - Cortica- Carlsbad, Carlsbad, California
  - Cortica- Glendale, Glendale, California
  - Cortica- Irvine, Irvine, California
  - Cortica- Laguna Niguel, Laguna Niguel, California
  - Cortica- San Diego, San Diego, California
  - Cortica- Marin, San Rafael, California
  - Cortica- Torrance, Torrance, California
  - Cortica- Westlake Village, Westlake Village, California
  - Cortica- Ridgefield, Ridgefield, Connecticut
  - Cortica- Trumbull, Trumbull, Connecticut
  - Cortica- Naperville, Naperville, Illinois
  - Cortica- Westchester, Westchester, Illinois
  - Cortica- Burlington, Burlington, Massachusetts
  - Cortica- Dedham, Dedham, Massachusetts
  - Cortica- Shrewsbury, Shrewsbury, Massachusetts
  - Cortica- Plano, Plano, Texas
  - Cortica- The Woodlands, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No
No plans to share